CLINICAL TRIAL: NCT00782704
Title: Development and Validation of a Morbidity Index for Complications in Minor and Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ksenija Slankamenac, MD PhD, University of Zurich
Other Study IDs: StV 30-2008
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Postoperative Complications
Keywords: A self-administered questionnaire to collect data from patients, physicians and nurses about the severity of postoperative surgical complications.; Based on this questionnaire we will develop the morbidity index
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: questionnair for Patients
- 2: questionnaire for Nurses
- 3: questionnaire for Physicians

SUMMARY:
The aim is to develop and validate a morbidity index for postoperative complications in patients undergoing visceral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Capacity to act and no legal guardian
* Patients with any underlying disease admitted to the Department of Visceral and Transplantation Surgery of the University Hospital of Zurich with planned minor or major visceral surgery
* German language as daily language.

Exclusion Criteria:

* Patients with cognitive difficulties and diseases, which may yield unreliable answers
* Patients unable to read and write

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients: all patients of the Department of Visceral and Transplantation Surgery of the University Hospital of Zurich Nurses: Staff nurses of the University Hospital of Zurich Physicians: from different units of the University Hospital of Zurich (Visceral-, Thoracic, Cardiovascular Surgery, Anesthesiology, Intensiv Care Unit, Urology)
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
to develop and validate a morbidity index | preoeprativ and one day before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ksenija Slankamenac, med. pract, Principal Investigator — Department of Visceral and Transplantation Surgery
Locations (1):
- Department of Visceral and Transplantation Surgery of the University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland